CLINICAL TRIAL: NCT03406364
Title: A Phase I Study to Assess the Safety and Activity of Combined MG005 and Sorafenib (NEXAVAR®) Treatment in Patients With Solid Tumor
Brief Title: Assess the Safety and Activity of Combined MG005 and Sorafenib (NEXAVAR®) Treatment With Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Metagone Biotech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MEOMG1A20170313
Record Dates: First submitted 2018-01-08; First posted 2018-01-23 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Solid Tumor

STUDY DESIGN:
Intervention Model Description: Phase I:
  Eligible subjects will receive 1 of 3 different dosages of the combination therapy of GW5074 and sorafenib. The dose cohorts include:
  * Monotherapy with 750 mg QD GW5074, followed by 750 mg QD GW5074 + 200 mg QD Sorafenib
  * 1500 mg QD GW5074 + 200 mg QD Sorafenib
  * 750 mg BID GW5074 + 200 mg QD Sorafenib
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MG005 (Experimental): Cohort 1 :3 × 250 mgMG005+1 × 200 mgSorafenib[8:00 AM (±2 hours)] Cohort 2 :6 × 250 mgMG005+1 × 200 mgSorafenib[8:00 AM (±2 hours)] Cohort 3 :3 × 250 mgMG005+1 × 200 mgSorafenib; 3 × 250 mgMG005+1 × 200 mgSorafenib[8:00 AM (±2 hours); 8:00 PM (±2 hours)]
  Interventions: Drug: MG005

INTERVENTIONS:
Drug: MG005 — Phase I:
  Eligible patients will receive different dosages of GW5074 in 1 of the 3 dose cohorts plus 200 mg of sorafenib. Dose cohorts will be escalated sequentially from Cohort 1 at 750 mg QD GW5074 plus 200 mg QD sorafenib to Cohort 2 at 1500 mg QD GW5074 plus 200 mg QD sorafenib, and Cohort 3 at 750 mg BID GW5074 plus 200 mg QD sorafenib. Owing to the fact that there is no previous human experience for GW5074, Cohort 1 will include a monotherapy stage with 750 mg QD GW5074 prior to administration of the GW5074 and sorafenib combination to initially assess the safety of GW5074 monotherapy.

SUMMARY:
The proposed initial trial is a Phase I, open label study to evaluate the safety and explore efficacy of MG005 in combination with sorafenib in patients with solid tumor. The eligible patients will receive 200 mg of sorafenib with 3 pre-defined dose levels of GW5074, escalated from 750 mg to 1500 mg (daily dose), to determine the Maximum Tolerated Dose (MTD) and dose limiting toxicities (DLT) (if any) at Phase I stage.

ELIGIBILITY:
Inclusion Criteria:

1. Patient who is able to understand the nature of this study and accepts to enter the study by signing written informed consent
2. Patients who are ≥ 20 years of age
3. Patients with histologically confirmed advanced or metastatic disease that is either refractory to or intolerant of existing standard therapy or for which no effective standard therapy that confers clinical benefit is available (patients may have received prior therapy with sorafenib if not intolerable)
4. Patient has at least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
5. Patient able to provide either an archived tumor sample or with accessible tumor for biopsy and willingness to provide it prior to initiation of study treatment
6. At least 4 weeks post any therapeutic modalities (e.g., surgery, radiotherapy, and therapeutic agents) prior to initial dosing except the palliative radiotherapy performed on non-study-related local lesions
7. Eastern Cooperative Oncology Group (ECOG) performance score ≤ 2 8.Patient's life expectancy of at least 3 months

9.Patient has adequate hematopoietic, hepatic function and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to screening:

* Hemoglobin ≥ 9.0 g/dL
* Absolute neutrophil count (ANC) ≥ 1,500 cells/μL
* Total white blood cell (WBC) ≥ 3,000 cells/μL
* Platelet ≥ 100,000 counts/μL
* Total bilirubin ≤ 1.5× upper limit of normal (ULN) and no sign of jaundice
* ALT and AST ≤ 2.5× ULN (≤ 5× ULN for patients with liver involvement)
* ALP ≤ 5× ULN
* Creatinine ≤ 1.5× ULN
* Potassium, total calcium and magnesium within normal limits or correctable with supplements 10.Patient is able to take food and drug orally. 11.Patient is able to correctly operate the provided digital sphygmomanometer. 12.Female patient with childbearing potential should be confirmed of not being pregnant or not lactating at the screening and during the study.

  13.Patient is willing to comply with protocol-stated requirements, instructions and restrictions.

Exclusion Criteria:

1. Patient who has participated in other investigational studies and received any investigational therapy within 4 weeks prior to study dosing
2. Patient carries history of primary malignancy other than the entry diagnosis except curatively treated non-melanoma skin cancer, cervical carcinoma in situ, or superficial bladder tumors within 5 years prior to study entry.
3. Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of GW5074 and sorafenib (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
4. Patient with known leptomeningeal or brain metastasis (including those who require glucocorticoids or intrathecal chemotherapy) by radiologic/histological evidence, or only bone metastasis
5. Patient with history of significant cardiac disease including superior vena cava, unstable angina, congestive heart failure > class 2 per New York Heart Association (NYHA) classification, cardiac arrhythmias, cardiac ischemia/infarction, long QT-syndrome (i.e., QTc > 450 msec for males and > 470 msec for females), poorly controlled hypertension (systolic blood pressure > 150 mm-Hg and/or diastolic blood pressure > 90 mm-Hg on anti-hypersensitive medications), and valvular heart disease
6. History of organ or bone marrow transplant
7. Patient who has not recovered from side/toxic effects of previous therapy (i.e., NCI-CTCAE grade 1 or less) prior to the first dose of study medications
8. Patients who are receiving or with conditions requiring substances that are potent inducers of CYP3A4 activity (e.g., rifampin, St. John's wort, phenytoin, carbamazepine, phenobarbital, and dexamethasone)
9. Patients who are receiving or with conditions requiring sensitive substrates of CYP1A2, 1B1, 2C8, 2C19 and 3A4 with narrow therapeutic windows (e.g., theophylline, duloxetine, alosetron, tizanidine, repaglinide, omeprazole, S-mephenytoin, alfentanil, sirolimus, pimozide, and tacrolimus)
10. History of stroke or transient ischemic attack within 6 months of study entry
11. Patient with any hemorrhage/bleeding event (e.g., non-healing wound, ulcer, and bone fracture) ≥ NCI-CTCAE grade 2 within 28 days prior to study treatment, or history of bleeding diathesis or coagulopathy
12. Patients with poorly controlled ascites and/or requirement for therapeutic paracentesis more frequently than once every 3 months
13. Patients with HIV, acute HBV, and HCV (except hepatitis carriers) infections
14. Patient with known or suspected hypersensitivity to any agent given in the course of this trial
15. Patient with underlying medical, mental or psychological conditions that would impair the treatment compliance, or in the opinion of the investigator would not permit to participate in the study
16. Male and female patients (with child-bearing potential [between puberty and 2 years after menopause]) who are unwilling to practice an effective method of birth control (safe hormonal methods or/and barrier contraception) during the entire study period and 2 months after the last study drug intake

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2020-01-09 (Actual); Study Completion 2020-07-24 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose(MTD)and Dose Limiting(DLT) -phase I | DLTs will be assessed during the initial 8-week treatment periods for Cohort 1.
  MTD by defining DLTs for MG005 and in combination with sorafenib.
Maximum Tolerated Dose(MTD)and Dose Limiting(DLT) -phase I | DLTs will be assessed during the initial 4-week treatment periods for Cohort 2/3
  MTD by defining DLTs for MG005 and in combination with sorafenib.

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-Service General Hospital, Taipei, Nehu District, Taiwan